CLINICAL TRIAL: NCT03535987
Title: Pilot Cohort Study of Rb-82 Myocardial PET Imaging to Evaluate Coronary Microvascular Dysfunction in Men With Prostate Cancer Receiving Androgen-Deprivation Therapy
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 18817
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Observational: To determine the feasibility of using myocardial PET imaging
  Interventions: Device: myocardial PET imaging

INTERVENTIONS:
Device: myocardial PET imaging — using myocardial PET imaging as a means to assess cardiovascular risk in men with prostate cancer planned for androgen-deprivation therapy with external beam radiation therapy

SUMMARY:
To determine the feasibility of using myocardial PET imaging as a means to assess cardiovascular risk in men with prostate cancer planned for androgen- deprivation therapy with external beam radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Either clinically localized prostate cancer or biochemically-recurrent prostate cancer patients who are planned for at least 6 months ADT with a GnRH agonist and curative-intent radiation therapy per their oncologic providers.
* Over 50 years of age. Calculated 10-year Framingham General Cardiovascular Risk Score of ≥10% at the time of planned initiation of ADT.
* Patients must be able to read and understand English.
* Participants must sign the informed consent form.

Exclusion Criteria:

* Prior treatment with GnRH agonist therapy.
* History of active asthma or other reactive airway disease.
* Ischemic cardiac event (myocardial infarction, unstable angina) within the preceding 6 months.

Min Age: 51 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — using myocardial PET imaging as a means to assess cardiovascular risk in men with prostate cancer planned for androgen-deprivation therapy with external beam radiation therapy
Study Population: men with clinically-localized or biochemically recurrent prostate cancer planned for curative-intent external beam radiation therapy with concomitant ADT for a duration of at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-10-19 (Actual)

PRIMARY OUTCOMES:
number of subjects who successfully complete Rb-82 myocardial PET Imaging assessments | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Narayan, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT03535987/ICF_000.pdf